CLINICAL TRIAL: NCT01921192
Title: Effect of Folic Acid, Vitamin B6 and Vitamin B12 in Diabetic Retinopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Mariano Malaguarnera, Associate Professor, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1/2012
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Non Proliferative Diabetic Retinopathy; Proliferative Diabetic Retinopathy
MeSH Terms: interventions — Folic Acid; Vitamin B 6; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Folic Acid, vit B6 and B12 (Active Comparator)
  Interventions: Drug: Folic Acid, vit B6 and B12
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Folic Acid, vit B6 and B12
  Arms: Folic Acid, vit B6 and B12
Drug: Placebo
  Arms: Sugar pill

SUMMARY:
Homocysteine, a well-known inducer of vascular endothelial cell damage has been associated with extracellular matrix changes. Many studies demonstrated that high levels of this aminoacid in diabetic patients increases significantly the risk of the development of this pathology. This study has been undertaken to investigate the role of homocysteine and its cofactors (folic acid, vitamin B6 and B12) during the progression of the diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients with proliferative and non proliferative retinopathy

Exclusion Criteria:

* Patients with chronic liver disease Patients with kidney disease.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
homocysteine | 12 months

SECONDARY OUTCOMES:
folic acid | 12 months

OTHER OUTCOMES:
vitamin B6 | 12 months
vitamin B12 | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Catania, Cannizzaro Hospital, Catania, Italy